CLINICAL TRIAL: NCT05445622
Title: Assessing Student Learning of Spinal Mobilization With Real-time Objective Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 174-19
Record Dates: First submitted 2022-02-14; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects were able to practice spinal manipulation using the Activ5 device (Activbody, San Diego, CA, USA) for real-time objective visual feedback during in class lecture and lab. Activ5 device has a built-in force sensor that can provide realtime objective visual feedback via a Bluetooth connected mobile device.
  Interventions: Other: learning spinal mobilization with a force sensor
- Control (Active Comparator): Subjects were taught spinal mobilization using the traditional approach.
  Interventions: Other: learning spinal mobilization with a force sensor

INTERVENTIONS:
Other: learning spinal mobilization with a force sensor — Experimental group will use a force sensor (Active5) while learning spinal mobilization during the practice lab portion of the class. The force sensor will provide objective feedback to the students. Each student will be instructed on how to use the Active 5 device prior to utilization it in the classroom setting.

SUMMARY:
This is a research project on physical therapy education. Subjects will be recruited using convenience sampling from second-year physical therapy students on the campus of Youngstown State University. There are currently 28 students in the class. All students will be recruited to participate in the study. The objective of the study is to assess student learning of grades of spinal mobilization with real-time objective feedback.

DETAILED DESCRIPTION:
Sampling: Subjects will be recruited using convenience sampling from second-year physical therapy students on the campus of Youngstown State University.

Research Design: Randomized controlled trial (RCT). Subjects will be randomly assigned to the experimental group or control group. Subjects will attend a spinal mobilization lecture followed by a practice lab.

Randomization: Once enrolled in the study, each student will be randomly assigned to experimental or control groups. Randomization will occur via a random number generator and allocation will be concealed in opaque envelopes.

Intervention:

The experimental group will use a force sensor (Active5) while learning spinal mobilization during the practice lab portion of the class. The force sensor will provide objective feedback to the students. Each student will be instructed on how to use the Active 5 device prior to utilizing it in the classroom setting. The device can display the amount of force generated by the student on a smartphone or a tablet in real-time so the students would be able to adjust the amount of force.

The Control group will participate in the same classroom lecture and activity. However, during the practice lab portion of the class, the control group will only receive traditional subjective feedback from the class instructor and/or student peers.

A perceived competence scale survey (score between 0-10 with 10 being confident and 0 being not confident) with demographic information will be administered immediately after the intervention. An independent blinded instructor will serve as the assessor of student skill level to avoid bias immediately after the intervention/procedure. Student t-test will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Second year Physical Therapy students; males or females; age between 20 and 60 years of age.

Exclusion Criteria:

* Student who is not a second year Physical Therapy student or unwilling to participate in the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
A perceived competence scale survey instructor will serve as the assessor of student skill level to avoid bias. Student t test will be used for data analysis. Perceived competence scale survey | immediately after the intervention/procedure
  A self reporting survey (score between 0-10 with 10 being confident and 0 being not confident)

SECONDARY OUTCOMES:
Student mobilization skill | immediately after the intervention/procedure
  Assessed by instructor on 0-10 scale (10 being a satisfactory and 0 being not satisfactory)

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Ge, DPT, PhD, Principal Investigator — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No